CLINICAL TRIAL: NCT06893029
Title: Visually Induced Dizziness in Concussed and Non-Concussed Dizzy Patients: Identifying the Pathophysiology of Postural Control Upon Optokinetic Stimuli
Brief Title: Dizziness Due to Visual Stimuli in Patients With Concussion and Other Causes of Dizziness: Examination of Balance Behaviour
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dominik Straumann (Other)
Collaborators: University Hospital, Zürich (Other); BrainCare Medical Group (Other)
Responsible Party: Sponsor-Investigator, Dominik Straumann, Prof. Dr. med., University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2024-00956
Record Dates: First submitted 2025-03-06; First posted 2025-03-25 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Dizziness; Concussion (Diagnosis); Traumatic Brain Injury; Balance Assessment
Keywords: Visually induced dizziness
MeSH Terms: conditions — Dizziness; Brain Concussion; Disease; Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: The project is organised in 4 arms, as healthy subjects and patients will be examined. Optokinetic stimulation will be applied to eighter by a physical disc or a head mounted device using virtual application. Healthy subjects will conduct a physical and a virtual balance assessment with visual stimulation, in a cross-over design. Patients will only conduct one type of balance assessment, physical or virtual, to prevent symptom exacerbation. This limitation for dizzy patients is based on the experience of leading clinicians from the vertigo center and on former research projects in the field of VID (de Vestel, et al., 2022; Guerraz et al., 2001; van Ombergen et al., 2016).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy Subjects (Physical / Virtual) (Active Comparator): Cross-over design for healthy subjects, physical optokinetic stimulation in advance to virtual optokinetic stimulation.
  Interventions: Diagnostic Test: Postural Response upon physical optokinetic stimulation; Diagnostic Test: Postural Response upon virtual optokinetic stimulation
- Healthy Subjects (Virtual / Physical) (Active Comparator): Cross-over design for healthy subjects, virtual optokinetic stimulation in advance to physical optokinetic stimulation.
  Interventions: Diagnostic Test: Postural Response upon physical optokinetic stimulation; Diagnostic Test: Postural Response upon virtual optokinetic stimulation
- Patients (Physical) (Experimental): These patients are only examined with the physical stimulation to avoid excessive symptom burden.
  Interventions: Diagnostic Test: Postural Response upon physical optokinetic stimulation
- Patients (Virtual) (Experimental): These patients are only examined with the virtual stimulation to avoid excessive symptom burden.
  Interventions: Diagnostic Test: Postural Response upon virtual optokinetic stimulation

INTERVENTIONS:
Diagnostic Test: Postural Response upon physical optokinetic stimulation — The physical optokinetic stimulation consists of rotating stimulation in either direction using a physical disc (de Vestel, et al., 2022; Guerraz et al., 2001; van Ombergen et al., 2016). The assessment is conducted in complete dark, unless the fluorescent dots (approx. 11% covered of the disc area.). The disc has a diameter of 1 m. Stimulation time per trial will be 30 s.
  Arms: Healthy Subjects (Physical / Virtual); Healthy Subjects (Virtual / Physical); Patients (Physical)
Diagnostic Test: Postural Response upon virtual optokinetic stimulation — The virtual optokinetic stimulation is implemented in virtual reality goggles (Meta Quest 3, Meta Platforms, Menlo Park, CA, USA) applying oscillating and rotating stimulation in frontal and vertical axis with coherent or incoherent stimuli. The assessment in the virtual environment will be as similar as possible compared the physical stimulation. Hence, the virtual environment simulation complete dark, unless the fluorescent dots (approx. 15% covered of the disc area.). In addition to the rotating condition, the virtual dots are able to oscillate on the horizontal or vertical axis to create a more sensitive evaluation method than the physical one (Laurens et al., 2011). Stimulation time per trial will be 30 s.
  Arms: Healthy Subjects (Physical / Virtual); Healthy Subjects (Virtual / Physical); Patients (Virtual)

SUMMARY:
This research project aims to measure how balance is affected by special visual stimulation. Dizziness caused by complex moving visual patterns, known as optokinetic stimulation, is usually called visually induced dizziness (VID).

The study includes patients with persistent symptoms after a concussion and those with non-traumatic dizziness. Healthy participants serve as a control group for the comparison of balance and symptom responses.

The optokinetic stimulation is done using either a physical rotating disk or a virtual reality (VR) headset. The visual effects are created by bright moving dots. During the stimulation, these patterns move in a specific manner and directions while the subject's balance is recorded. Symptoms such as dizziness, headache, and nausea are also documented.

The goal of this project is to improve objective diagnosis of VID. By comparing patients and healthy subjects, the study aim to assess the severity of the disorder. It is also assumed that using different visual stimuli during the balance assessment will offer more sensitive and accurate results.

In the long term, this innovative assessment method shall support clinicians to establish the diagnosis of VID, and improve the treatment and management of patients with VID.

DETAILED DESCRIPTION:
Sport-related concussion (SRC) refers to traumatic head injuries caused by direct biomechanical forces to the head, neck or body during physical activity. Due to very heterogeneous clinical patterns in concussed patients including multiple clinical profiles and subtypes, standardised diagnosis for SRC is still in scope of research. Thus, diagnostic procedures are currently based on clinical examination and subjective complaints using questionnaires, while objective assessments supporting a diagnosis for concussed patients are lacking. Only some functional limitations are recorded via objective methods, but no quantification and no diagnosis are possible.

Common questionnaires to assess VID in concussed patients and for vestibular disorders are the visual vertigo analogue scale (VVAS), and the situational vertigo questionnaire (SVQ), though there exist more. The dizziness handicap inventory (DHI) is used to classify the general aspect of dizziness. Other methods to support VID diagnosis have been developed including subjective visual vertical assessment or balance screenings with optokinetic stimulation. Such objective findings are essential for a reliable diagnosis supporting subjective complaints. However, determined parameters and observed pathologies vary among studies and thus, a classification via objective assessments in VID patients is still in scope of research. Nevertheless, symptom assessment is still considered as one of the best and reliable method to support diagnosis and success in treatment.

Outcomes of previously discussed and used questionnaires to assess VID rely on patients' compliance. Subjective evaluations on dizziness are challenging for patients and may therefore diverge from objective measurements. In addition, questionnaires do not explicitly distinguish between vertigo and dizziness. Moreover, self-reported symptoms showed moderate correlation to objective findings. This highlights the importance of realising objective methods such as balance assessments.

Some objective assessments to identify VID, and to discriminate among patient groups and healthy subjects have been introduced. But most of the studies investigating VID examined a broad variety of vestibular disorders, rarely including concussion.

Concerning balance assessment combined with optokinetic stimulation, several studies found significant differences among control groups and patients with vestibular disorders and dizziness, but findings varied across calculated parameters. Overall, mean deviations on sway path tended to be more predictive than lean sway, and significant effects are supposed to be in stimulated planes. Additionally for path length, there exists two quotients representing the balance response ratio between eyes open and eyes closed (Romberg quotient), and the ratio between eyes open and optokinetic stimulation (optokinetic quotient), which both showed significant effects comparing healthy subjects and visual vertigo patients. However, parameters evaluated from velocity were often in favour compared to path length. Furthermore, prolonged exposure to optokinetic stimulation triggered symptoms in patients with visual vestibular mismatch but not in control subjects, supporting the hypotheses of symptom exacerbation by visual motion. Regarding defined triggers for VID, one could assume that triggers are based on an individual level and therefore include various visual motion conditions such as complex, large-field or moving elements in order to conflict one's sensory integration. Given those multidimensional conditions for an assessment, the use of VR environments for this project benefits a broad and flexible range in VID assessment. Regarding the mentioned studies, one could assume that balance evaluation on multiple optokinetic stimuli and comparison to reference values based on healthy subjects has the potential to increase the sensitivity of the balance screening for VID subjects, and in particular concussed patients.

This project aims to generate greater reliability using a more differentiated balance assessment with optokinetic stimulation. Findings are assumed to help identifying potential VID on a more individual basis and support accurate classification.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years
* Binocular vision
* Recent concussion/mTBI within 4 weeks to 18 months post-injury for concussed patients
* Diagnosis related to dizziness or VID within 4 weeks to 18 months for non-concussed dizzy patients (including vestibular migraine)
* Signed ICF for included participants or signed general consent for retrospectively included patients if an ICF cannot be obtained.

Exclusion Criteria:

* BMI greater than 30
* Acute vestibular syndrome lasting at least 24 hours
* Severe non-correctable visual impairment
* Balance issues not dizziness-related, including:

  1. Neurological conditions (e.g., migraine)
  2. Orthopaedic conditions (e.g., lower extremity injury)
  3. Infectious diseases
  4. Other medical contexts
* Dizziness attributed to prescribed drugs, substance abuse, or mental disorders
* Cognitive impairments compromising task comprehension
* Preceding history of traumatic brain injury in the last 12 months
* History of severe traumatic brain injury with persisting impairments
* Other potentially confounding problems (e.g., psychiatric disease)
* Frequent episodes of rotatory vertigo

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of Postural Response to Optokinetic Stimulation | Time Point 1: During the first intervention, measurement on a single day. Time Point 2: 15 minutes after the first intervention, measurement on a single day
  To identify visually induced dizziness through the balance assessment, cutoff values based on calculated balance parameters will be evaluated to differentiate balance responses between concussed patients, non-concussed dizzy patients, and healthy controls. The reference will be the VID assessment performed during the clinical examination.
  Measurement Tool:
  * 6D sensor system (accelerometer and gyroscope) placed on the lower back and head.
  * acceleration in m/s^2
  * gyroscope in deg/s)
  Unit of Measure: Calculations on the balance responses from each measuring site and sensor type (accelerometer, gyroscope) include temporal and spectral parameters such as:
  * 95% area of motion (m^2/s^4, deg^2/s^2)
  * RMS, SD, Mean (m/s^2, deg/s)
  * Power Spectral Density (PSD) between 0.1-2 Hz ((m^2/s^4)/Hz, (deg^2 /s^2)/Hz)
  * Power Spectral Density (PSD) at stimulation frequency of 1/3 Hz((m^2/s^4)/Hz, (deg^2 /s^2)/Hz)
  Comparison:
  * Balance parameters among the investigated groups

SECONDARY OUTCOMES:
Identification of Different Postural Characteristics Response to Optokinetic Stimulation | Time Point 1: During the first intervention, measurement on a single day. Time Point 2: 15 minutes after the first intervention, measurement on a single day
  It is hypothesized that patients with different diagnoses will exhibit distinct postural response patterns, which can be quantified and categorised. Based on the diagnosis, specific characteristics from the determined parameters shall be analysed.
  Measurement Tool:
  * 6D sensor system (accelerometer and gyroscope) placed on the lower back and head.
  * acceleration in m/s^2
  * gyroscope in deg/s)
  Unit of Measure: Calculations on the balance responses from each measuring site and sensor type (accelerometer, gyroscope) include temporal and spectral parameters such as:
  * 95% area of motion (m^2/s^4, deg^2/s^2)
  * RMS, SD, Mean (m/s^2, deg/s)
  * Power Spectral Density (PSD) between 0.1-2 Hz ((m^2/s^4)/Hz, (deg^2 /s^2)/Hz)
  * Power Spectral Density (PSD) at stimulation frequency of 1/3 Hz((m^2/s^4)/Hz, (deg^2 /s^2)/Hz)
  Comparison:
  * Differences and rates of change in determined parameters are clustered across these groups
Severity of Visually Induced Dizziness | Time Point 1: During the first intervention, measurement on a single day. Time Point 2: 15 minutes after the first intervention, measurement on a single day
  The balance assessment outcome shall be used to categorise the severity of visually induced dizziness based on calculated balance parameters.
  Measurement Tool:
  * 6D sensor system (accelerometer and gyroscope) placed on the lower back and head.
  * acceleration in m/s^2
  * gyroscope in deg/s)
  Unit of Measure: Calculations on the balance responses from each measuring site and sensor type (accelerometer, gyroscope) include temporal and spectral parameters such as:
  * 95% area of motion (m^2/s^4, deg^2/s^2)
  * RMS, SD, Mean (m/s^2, deg/s)
  * Power Spectral Density (PSD) between 0.1-2 Hz ((m^2/s^4)/Hz, (deg^2 /s^2)/Hz)
  * Power Spectral Density (PSD) at stimulation frequency of 1/3 Hz((m^2/s^4)/Hz, (deg^2 /s^2)/Hz)
  Comparison:
  * Balance parameters will be classified into clusters, such as normal, borderline, and abnormal balance behaviour.

OTHER OUTCOMES:
Comparison of virtual and physical optokinetic stimulation in healthy subjects | Time Point 1: During the first intervention, measurement on a single day. Time Point 2: 15 minutes after the first intervention, measurement on a single day
  Balance responses will be compared between the two arms of healthy subjects who complete both types of balance assessments (virtual and physical optokinetic stimulation).
  Measurement Tool:
  * 6D sensor system (accelerometer and gyroscope) placed on the lower back and head.
  * acceleration in m/s^2
  * gyroscope in deg/s)
  Unit of Measure: Calculations on the balance responses from each measuring site and sensor type (accelerometer, gyroscope) include temporal and spectral parameters such as:
  * 95% area of motion (m^2/s^4, deg^2/s^2)
  * RMS, SD, Mean (m/s^2, deg/s)
  * Power Spectral Density (PSD) between 0.1-2 Hz ((m^2/s^4)/Hz, (deg^2 /s^2)/Hz)
  * Power Spectral Density (PSD) at stimulation frequency of 1/3 Hz((m^2/s^4)/Hz, (deg^2 /s^2)/Hz)
  Comparison:
  * Balance parameters among healthy controls.

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - BrainCare Medical Group, Zurich, Canton of Zurich
  - University Hospital Zurich, Department of Neurology, Zurich, Canton of Zurich

IPD SHARING:
Plan to Share IPD: Yes
Data from the CRF, raw values from the balance measurements, and calculated balance parameter will be shared IPD:
  * Diagnosis related to VID:
  * Group assignment
  * Informed Consent
  * Anthropometric data (weight, height)
  * Age
  * Questionnaire's data: DHI, VVAS, SVQ, SSQ
  * Symptom burden during balance assessment
  * Completion of assessment
  * Balance raw data
  * Calculated balance parameters
Time Frame: 01.01.2026 (before publication) - 01.01.2030 (3 years after publication)
Access Criteria: Associates from the University of Zurich: Full access to anonymised IPD Access to IPD and supporting information will be granted to other researchers and reviews who first establish contact with the Sponsor of University of Zurich and provide a detailed description of their research plan. Upon approval, data will be shared through a secure access system in compliance with institutional and ethical guidelines.

REFERENCES:
- [Background] Laurens J, Awai L, Bockisch CJ, Hegemann S, van Hedel HJ, Dietz V, Straumann D. Visual contribution to postural stability: Interaction between target fixation or tracking and static or dynamic large-field stimulus. Gait Posture. 2010 Jan;31(1):37-41. doi: 10.1016/j.gaitpost.2009.08.241. Epub 2009 Sep 22. PMID 19775892
- [Background] Agarwal K, Bronstein AM, Faldon ME, Mandala M, Murray K, Silove Y. Visual dependence and BPPV. J Neurol. 2012 Jun;259(6):1117-24. doi: 10.1007/s00415-011-6311-7. Epub 2011 Nov 24. PMID 22113702
- [Background] Fife TD, Giza C. Posttraumatic vertigo and dizziness. Semin Neurol. 2013 Jul;33(3):238-43. doi: 10.1055/s-0033-1354599. Epub 2013 Sep 21. PMID 24057827
- [Background] Bisdorff AR, Staab JP, Newman-Toker DE. Overview of the International Classification of Vestibular Disorders. Neurol Clin. 2015 Aug;33(3):541-50, vii. doi: 10.1016/j.ncl.2015.04.010. PMID 26231270
- [Background] Kontos AP, Sufrinko A, Sandel N, Emami K, Collins MW. Sport-related Concussion Clinical Profiles: Clinical Characteristics, Targeted Treatments, and Preliminary Evidence. Curr Sports Med Rep. 2019 Mar;18(3):82-92. doi: 10.1249/JSR.0000000000000573. PMID 30855306
- [Background] Van Ombergen A, Lubeck AJ, Van Rompaey V, Maes LK, Stins JF, Van de Heyning PH, Wuyts FL, Bos JE. The Effect of Optokinetic Stimulation on Perceptual and Postural Symptoms in Visual Vestibular Mismatch Patients. PLoS One. 2016 Apr 29;11(4):e0154528. doi: 10.1371/journal.pone.0154528. eCollection 2016. PMID 27128970
- [Background] Pavlou M, Davies RA, Bronstein AM. The assessment of increased sensitivity to visual stimuli in patients with chronic dizziness. J Vestib Res. 2006;16(4-5):223-31. PMID 17538212
- [Background] Patricios JS, Schneider KJ, Dvorak J, Ahmed OH, Blauwet C, Cantu RC, Davis GA, Echemendia RJ, Makdissi M, McNamee M, Broglio S, Emery CA, Feddermann-Demont N, Fuller GW, Giza CC, Guskiewicz KM, Hainline B, Iverson GL, Kutcher JS, Leddy JJ, Maddocks D, Manley G, McCrea M, Purcell LK, Putukian M, Sato H, Tuominen MP, Turner M, Yeates KO, Herring SA, Meeuwisse W. Consensus statement on concussion in sport: the 6th International Conference on Concussion in Sport-Amsterdam, October 2022. Br J Sports Med. 2023 Jun;57(11):695-711. doi: 10.1136/bjsports-2023-106898. PMID 37316210
- [Background] Guerraz M, Yardley L, Bertholon P, Pollak L, Rudge P, Gresty MA, Bronstein AM. Visual vertigo: symptom assessment, spatial orientation and postural control. Brain. 2001 Aug;124(Pt 8):1646-56. doi: 10.1093/brain/124.8.1646. PMID 11459755
- [Background] De Vestel C, De Hertogh W, Van Rompaey V, Vereeck L. Comparison of Clinical Balance and Visual Dependence Tests in Patients With Chronic Dizziness With and Without Persistent Postural-Perceptual Dizziness: A Cross-Sectional Study. Front Neurol. 2022 May 24;13:880714. doi: 10.3389/fneur.2022.880714. eCollection 2022. PMID 35685740
- [Background] Dannenbaum E, Chilingaryan G, Fung J. Visual vertigo analogue scale: an assessment questionnaire for visual vertigo. J Vestib Res. 2011;21(3):153-9. doi: 10.3233/VES-2011-0412. PMID 21558640